CLINICAL TRIAL: NCT00879229
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Parallel-Group Study to Evaluate the Efficacy and Safety of Ambrisentan in Subjects With Idiopathic Pulmonary Fibrosis and Pulmonary Hypertension
Brief Title: ARTEMIS-PH - Study of Ambrisentan in Subjects With Pulmonary Hypertension Associated With Idiopathic Pulmonary Fibrosis
Acronym: ARTEMIS-PH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-300-0128
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2014-04-22 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Idiopathic Pulmonary Fibrosis; Pulmonary Hypertension
Keywords: Idiopathic Pulmonary Fibrosis; Pulmonary Hypertension; PH; IPF; Ambrisentan; ERA; Endothelin Receptor Antagonist; Cardiovascular
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Hypertension, Pulmonary | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambrisentan (Experimental): Participants were randomized to receive ambrisentan treatment at an initial dose of 5 mg for 4 weeks, followed by ambrisentan at the target dose of 10 mg for an additional 52 weeks
  Interventions: Drug: Ambrisentan
- Placebo (Placebo Comparator): Participants were randomized to receive placebo to match ambrisentan for 48 weeks, then transition to ambrisentan treatment at the initial dose of 5 mg for 4 weeks, followed by ambrisentan at the target dose of 10 mg for an additional 4 weeks.
  Interventions: Drug: Ambrisentan; Drug: Placebo

INTERVENTIONS:
Drug: Ambrisentan — Ambrisentan (5 mg or 10 mg tablet) administered orally once daily.
  Other Names: Letairis
Drug: Placebo — Placebo to match ambrisentan administered orally once daily.
  Arms: Placebo

SUMMARY:
Ambrisentan is an endothelin receptor antagonist used for the treatment of pulmonary hypertension (PH). Based on research suggesting a role for endothelin-1 in the pathogenesis of idiopathic pulmonary fibrosis (IPF) and the poor prognosis for patients with IPF who are also diagnosed with PH, this study was designed to evaluate the effectiveness and safety of ambrisentan in that patient population.

ELIGIBILITY:
Selected Inclusion Criteria:

* Weight ≥ 40 kg at screening
* Diagnosis of IPF based on modified American Thoracic Society-European Respiratory Society guidelines
* Diagnosis of PH based on the following hemodynamic requirements: mean pulmonary artery pressure (mPAP ≥ 25 mm Hg; pulmonary vascular resistance > 240 dyne.sec/cm^5; pulmonary capillary wedge pressure or left ventricular end-diastolic pressure ≤ 15 mm Hg
* Forced vital capacity (FVC) ≥ 40%
* Able to walk at least 50 meters during two 6-minute walk tests
* If receiving calcium channel blockers, low-dose oral corticosteroids, immunosuppressive, cytoxic, or antifibrotic drugs dose must have been stable.

Selected Exclusion Criteria:

* Diagnosis of PH primarily due to an etiology other than IPF
* Surgical lung biopsy diagnosis other than Usual Interstitial Pneumonia
* Other known cause of interstitial lung disease
* Evidence of significant obstructive lung disease
* Recent hospitalization for an acute exacerbation of IPF
* Recent active pulmonary or upper respiratory tract infection
* Left ventricular ejection fraction < 40%
* Serum creatinine ≥ 2.5 mg/dL
* Required hemodialysis, peritoneal dialysis, or hemofiltration
* Female subject who was pregnant or breastfeeding
* Recent treatment for PH with an endothelin receptor antagonist (ERA), phosphodiesterase type 5 inhibitor, or prostacyclin derivative
* Recent treatment with high dose oral corticosteroids
* Recent treatment (within 4 weeks prior to screening) with imatinib mesylate (Gleevec)
* Alanine aminotransferase or aspartate aminotransferase lab value that was greater than 1.5 x the upper limit of the normal range
* Discontinued other ERA treatment for any adverse reaction other than those associated with liver function test abnormalities

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Gillies, M.D., Study Director — Gilead Sciences
Locations (85):
- United States (51):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California Davis, Davis, California
  - David Geffen School of Medicine UCLA, Los Angeles, California
  - University of California San Diego Medical Center, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Heatlh Sciences Center, Aurora, Colorado
  - Bay Area Chest Physicians, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami Medical Center, Miami, Florida
  - Suncoast Lung Center, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Atlanta Institute for Medical Research, Decatur, Georgia
  - University of Chicago, Chicago, Illinois
  - Kentuckiana Pulmonary Association, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deacones Medical Center, Boston, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Creighton University Center for Allergy & Asthma, Omaha, Nebraska
  - Dartmouth Medical School, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - Winthrop University Hospital, Mineola, New York
  - North Shore Health System, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland Case Western, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Alleghany General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Heart Institiute and Vascular Institute, Falls Church, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Providence Everett Medical Center, Everett, Washington
- Australia (3):
  - St. Vincents Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Perth Hospital, Perth, Western Australia
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Universitatsklinikum Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
- Canada (7):
  - Peter Loughheed Center- Calgary General Hospital, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier De L'Universite de Montreal, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Center, Montreal, Quebec
  - Centre de Pneumologie de L'Hospital Laval, Sainte-Foy, Quebec
- Germany (8):
  - Evangelische Lungenklinik Berlin, Berlin
  - Charite-Universitatsmedizin Berlin, Berlin
  - Krankenhaus Donaustauf der LVA, Donaustauf
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitat Greifswald, Greifswald
  - Medizinische Hochschule Hannover, Hanover
  - Thorax Klinik, Heidelberg
  - LMU Klinikum der Universitat, München
- Italy (9):
  - Azienda Ospedaliero Universitaria, Catania
  - Presidio Ospedaliero G.B. Morgagni, Forlì
  - Ospedale S.Giuseppe Fatebenefratelli, Milan
  - Unita Funzionale di Pneumologia e Fisiopatologia Respiratoria, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Instituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione, Palermo
  - Policlinico Universitario Tor Vergata, Rome
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Centro delle Interstiziopatie Polmonari e Malattie Rare del Polmone, Torino
- United Kingdom (4):
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - University Hospital Aintree, Liverpool
  - University College Hosptial, London
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Ruocco G, Cekorja B, Rottoli P, Refini RM, Pellegrini M, Di Tommaso C, Del Castillo G, Franci B, Nuti R, Palazzuoli A. Role of BNP and echo measurement for pulmonary hypertension recognition in patients with interstitial lung disease: An algorithm application model. Respir Med. 2015 Mar;109(3):406-15. doi: 10.1016/j.rmed.2014.12.011. Epub 2015 Jan 3. PMID 25613108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in a total of 29 study sites in Australia, Europe, and North America. The first participant was screened on 21 October 2009. The last participant observation was on 22 February 2011.
Pre-assignment Details: 96 participants were screened; 40 participants were randomized and treated, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- Ambrisentan: Participants were randomized to receive ambrisentan treatment for 56 weeks
- Placebo: Participants were randomized to receive placebo for 48 weeks, followed by ambrisentan treatment for 8 weeks.
Period: Overall Study
Arm/Group | Ambrisentan | Placebo
Started | 25 | 15
Completed | 3 | 1
Not Completed | 22 | 14
Not completed — Study terminated by Sponsor | 13 | 12
Not completed — Death | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Clinical status did not improve | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants who were randomized and received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan | Placebo | Total
Number analyzed (Participants) | 25 | 15 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (7.7) | 68 (5.2) | 68 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 20 | 10 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 14 | 39
  Asian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 9 | 23
  Australia | 3 | 2 | 5
  Italy | 4 | 1 | 5
  Canada | 3 | 1 | 4
  Germany | 1 | 2 | 3
Baseline Dyspnea Index (BDI) [Mean (Standard Deviation); unit: units on a scale] — BDI range is 0 to 12 (worst to best).
  units on a scale | 5.0 (2.15) | 4.4 (2.10) | 4.8 (2.13)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Six-minute Walk Distance (6MWD).
Description: The change from baseline in 6MWD at Week 16 (end of blinded treatment) was evaluated.
Time Frame: Baseline to Week 16
Population: Participants in the Full Analysis Set (randomized and received at least one dose of study medication) with evaluable data were analyzed.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 21 | 9
meters | -96 (38) | -67 (51)
Statistical Analysis 1: Comparison: Ambrisentan vs Placebo; Test type: Superiority or Other; p = 0.696, Wilcoxon (Mann-Whitney) — This is an exact Wilcoxon rank sum test p-value for testing equality of ambrisentan and placebo distributions; Mean Difference (Final Values) = -29, 95% CI 2-sided [-54 to 17], Standard Error of Mean 67

2. Secondary Outcome: Long-term Survival
Description: Long-term survival was assessed as a Kaplan-Meier (KM) estimate of the percent probability of survival, with censoring at Week 48.
Time Frame: Week 48
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percent probability (KM% estimate)
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 25 | 15
percent probability (KM% estimate) | 22 [2.6 to 41.0] | 23 [0.0 to 52.5]

3. Secondary Outcome: Transition Dyspnea Index (TDI)
Description: The change in TDI at Week 16 (end of blinded treatment) was evaluated. TDI measures the change from the baseline characteristic "Baseline Dyspnea Index." The TDI range is -9 to +9 (worst to best; 0 = no change).
Time Frame: Baseline to Week 16
Population: Participants in the Full Analysis Set with evaluable data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 14 | 8
units on a scale | -1.5 (3.08) | -1.4 (3.78)

4. Secondary Outcome: Change From Baseline in WHO Functional Class
Description: WHO functional class rates severity of pulmonary hypertension, with 4 categories on a scale of 1 to 4 with the worst category being 4. Change is represented as an increase ("+1: Improved"), decrease ("-1: Deteriorated"), or no change ("0: No change") on the scale.
Time Frame: Baseline to Week 16
Population: Participants in the Full Analysis Set with evaluable data were analyzed.
Measure: Number; unit: units on a scale
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 14 | 8
units on a scale
  -1: Deteriorated | 0 | 1
  0: No change | 11 | 5
  +1: Improved | 3 | 2

5. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Percent Predicted
Description: FVC is a pulmonary function test, and is defined as the volume of air that can forcibly be blown out after taking a full breath. FVC% predicted is defined as FVC% of the patient divided by the average FVC% in the population for any person of similar age, sex and body composition.
Time Frame: Baseline to Week 16
Population: Insufficient data due to study termination
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP)
Description: Assessment of the the level of the amino acid fragment NT-proBNP is used to establish prognosis in cardiovascular disease.
Time Frame: Baseline to Week 16
Population: Insufficient data due to study termination
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in the Borg Dyspnea Index (BORG) Immediately Following Exercise
Description: Borg Dyspnea Index is a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness).
Time Frame: Baseline to Week 16
Population: Insufficient data due to study termination
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Hemoglobin-corrected Diffusing Capacity for Carbon Monoxide (DLCO) Percent Predicted
Description: DLCO is a pulmonary function test, and measures the partial pressure difference between inspired and expired carbon monoxide. DLCO% predicted is defined as DLCO% of the patient divided by the average DLCO% in the population for any person of similar age, sex and body composition.
Time Frame: Baseline to Week 16
Population: Insufficient data due to study termination
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Quality of Life (QOL) Score as Assessed by the Short-Form 36® (SF-36)
Description: Each SF-36 score is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. An increase in score indicates an improvement in health state.
Time Frame: Baseline to Week 16
Population: Insufficient data due to study termination
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in QOL Score as Assessed by the St. George's Respiratory Questionnaire (SRGQ)
Description: The SRGQ is designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Patients respond to questions about symptoms (frequency & severity) and impact components (social functioning and psychological disturbances resulting from airways disease). Scores range from 0 to 100, with higher scores indicating more limitations.
Time Frame: Baseline to Week 16
Population: Insufficient data due to study termination
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment
Description: Adverse events were collected based on the randomization group and not with regards to the specific treatment received.
Arm/Group | Ambrisentan | Placebo
Serious Adverse Events (participants affected / at risk) | 12/25 | 3/15
Other Adverse Events (participants affected / at risk) | 18/25 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=25) | Placebo (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=25) | Placebo (N=15)
Constipation (Gastrointestinal disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 5 | 3
Pyrexia (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Viral infection (Infections and infestations) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Cardiac murmur (Investigations) | 2 | 0
Eosinophil count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 3
Dizziness (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 2
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study GS-US-300-0128 was terminated early with enrollment of 40 of 225 planned subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years